CLINICAL TRIAL: NCT00043407
Title: A Phase I/II, Open Label, Multi-Center Study For The Evaluation Of CPG 7909 In Patients With Stage Iv Renal Cell Carcinoma
Brief Title: CPG 7909 in Patients Wih Stage IV Renal Cell Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C010; CO10, A8501022
Record Dates: First submitted 2002-08-08; First posted 2002-08-12 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal Cell Carcinoma, Phase I, Phase II, Immunotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPG 7909 Injection (Experimental)
  Interventions: Drug: CPG 7909

INTERVENTIONS:
Drug: CPG 7909 — In the phase I portion of the protocol, patients will be included in escalating dose groups: 0.08, 0.12, 0.16, 0.36, 0.54 or 0.81 mg/kg of CPG 7909 Injection. Patients will be treated once weekly subcutaneously for 24 weeks. In the Phase II portion of the trial patients will be treated at the MTD or the highest dose of 0.81 mg/kg identified in the Phase I dose escalation portion of the trial. All patients in Phase I and Phase II will be treated until disease progression or a maximum of 24 weeks.
  Other Names: PF-03512676

SUMMARY:
CPG 7909 given alone to patients with renal cell cancer after their nephrectomy. CPG 7909 is as a subcutaneous injection once per week for up to 24 weeks. Up to 40 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

Stage IV Renal Cell Carcinoma with lung and/or soft tissue metastasis Nephrectomy Measurable disease by RECIST criteria

Exclusion Criteria:

CNS, bone or Liver metastasis Tumors that are mainly papillary, chromophobe, medullary, collecting duct, or unclassified Prior immunotherapy, including IL-2 or IFN-alpha

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2002-03; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
To determine the tolerability of escalating doses of subcutaneously administered CPG 7909 Injection up to a maximum dose of 0.81 mg/kg in patients with metastatic renal cell cancer. | Indeterminate
To establish the maximum tolerated dose for CPG 7909 Injection as monotherapy in patients with metastatic renal cell cancer up to a dose of 0.81mg/kg. | Indeterminate
To estimate the overall tumor response rate of CpG 7909 according to the RECIST criteria in patients with metastatic renal cell cancer. | Indeterminate

SECONDARY OUTCOMES:
To assess tolerability relative to dose exposure, immunologic activity, the pharmacokinetic and pharmacodynamic profile of CPG 7909 Injection, time to progression, duration of response, and time to survival. | Indeterminate

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=CO10&StudyName=CPG%207909%20in%20Patients%20wih%20Stage%20IV%20Renal%20Cell%20Cancer